CLINICAL TRIAL: NCT00260494
Title: Acupuncture and Post-Surgical Wound Healing in Coronary Artery Bypass Graft Patients Undergoing Open Saphenous Vein Graft Harvest
Brief Title: Acupuncture and Post-Surgical Wound Healing
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: No difference in primary outcomes at interim analysis.
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: H7546-25444
Record Dates: First submitted 2005-11-29; First posted 2005-12-01 (Estimated); Last update posted 2013-07-23 (Estimated); Status verified 2013-07

CONDITIONS: Postoperative Complications; Surgical Wound Infection; Surgical Wound Dehiscence
Keywords: Cardiac Surgical Procedures; open saphenous vein graft harvest wounds; Postoperative Complications; Surgical Wound Infection; Surgical Wound Dehiscence
MeSH Terms: conditions — Postoperative Complications; Surgical Wound Infection; Surgical Wound Dehiscence | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- acupuncture (Experimental): acupuncture to lower extremity postoperatively
  Interventions: Other: acupuncture
- sham acupuncture (Sham Comparator): sham acupuncture at same sites.
  Interventions: Other: sham acupuncture
- control (No Intervention): no acupuncture, otherwise the same care and measurements

INTERVENTIONS:
Other: acupuncture — standardized acupuncture intended to improve blood flow and reduce edema to lower extremity.
  Arms: acupuncture
Other: sham acupuncture — standardized sham acupuncture at same sites as acupuncture.
  Arms: sham acupuncture

SUMMARY:
The purpose of this study is to determine if acupuncture improves wound healing. Since we, the investigators at the University of California, San Francisco (UCSF), know that how much oxygen is delivered to tissue is the best predictor of how well a wound will heal, we are measuring changes in tissue oxygen of wounds before and after acupuncture treatments. We are focusing on the leg wounds of coronary artery bypass graft (CABG) patients who have their saphenous veins harvested in an open fashion since this is a fairly well controlled patient model.

DETAILED DESCRIPTION:
This is a prospective, randomized, controlled pilot study of the effects of acupuncture on surgical site complications in patients undergoing coronary artery bypass grafting. The past forty years of research in the UCSF Wound Healing Laboratory have solidified the following observations:

1. without adequate oxygen delivery, many processes of wound healing cannot proceed normally, particularly resistance to infection, collagen deposition, angiogenesis, and inflammation; and
2. hypoxic conditions, unfortunately, are common in chronic and acute wounds, and often result from subcutaneous vasoconstriction.

Sympathetic nervous system (SNS) activators and other vasoconstrictors have been shown to produce wound hypoxia. Activation of the SNS by any means, including pain and anxiety, causes vasoconstriction and impairs oxygen delivery. Simple means that limit SNS activity have been shown to increase perfusion and oxygen tension, and thereby facilitate wound healing. Many preliminary studies have shown that acupuncture decreases SNS activation, pain, and anxiety. In addition, there is evidence that acupuncture enhances circulation of blood. We therefore hypothesize that acupuncture will facilitate wound healing. We aim to quantify changes in anxiety, pain, stress hormones, and perfusion and oxygenation induced by these interventions, as well as wound healing outcomes, including infection and other wound complications.

ELIGIBILITY:
Inclusion Criteria:

* Adults (age > 18)
* Males/females
* All races
* Elective/urgent CABG
* Open saphenous vein graft harvest
* University of California, San Francisco, and additional approved hospital sites

Exclusion Criteria:

Pre-operative

* Emergent CABG, valves
* History of peripheral vascular surgery, amputation, severe peripheral neuropathy, immunocompromise, or end-stage renal disease requiring hemodialysis

Post-operative

* Postoperative day 1 (POD1) hemodynamic instability
* ≥ 4u packed red blood cells transfusion (PRBC)/8 hours, CT > 200cc/hour 3 hours, > 2 pressors
* Prolonged intubation (> POD1)
* Altered mental status

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2005-03; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Transcutaneous tissue oxygen tension | postoperative days 0, 1, 2, 3

SECONDARY OUTCOMES:
ASEPSIS score | postoperatively
Transcutaneous tissue microperfusion | postoperative day 0, 1, 2, 3
Pain visual analogue scale (VAS) | postoperative days 0, 1, 2, 3
24-hour narcotic usage | postoperative days 0, 1, 2, 3
Anxiety VAS | postoperative days 0, 1, 2, 3
State-Trait Anxiety Inventory (STAI) | preoperative and postoperative
Serum epinephrine | postoperative
Serum cortisol | postoperative
Traditional Chinese Medicine pulse and tongue assessment | postoperative
Patient belief and expectancy survey | preoperative

OTHER OUTCOMES:
complications of acupuncture | duration of study

CONTACTS AND LOCATIONS:
Overall Officials: Harriet W Hopf, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States